CLINICAL TRIAL: NCT05494801
Title: Natural History, Disease Progression, and Long-Term Neurologic Sequelae of Ebola Virus Disease Survivors in PREVAIL III
Brief Title: Natural History, Disease Progression, and Long-Term Neurologic Sequelae of Ebola Virus Disease (EVD) Survivors in PREVAIL III
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000727; 000727-I
Record Dates: First submitted 2022-08-09; First posted 2022-08-10 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Ebola Virus Disease
Keywords: Emerging Infectious Disease; Hemorrhagic Fever; NEUROLOGIC SEQUELAE; Natural History
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; Communicable Diseases, Emerging; Hemorrhagic Fevers, Viral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Close Contacts: Close Contacts of EVD survivors, who were also previously in the PREVAIL III Neurology Substudy
- Patients (EVD Survivors): Participants with a history of Ebola Virus Disease who were involved in the Neurology Substudy of the PREVAIL III Ebola Natural History Study

SUMMARY:
Background:

Ebola virus disease (EVD) is a viral fever that can cause internal bleeding. The death rate from EVD is very high. In a 2014 outbreak in West Africa, 28,000 were affected and 11,000 died. EVD may also affect the brain and nervous system, but this is not well studied. People with EVD report headaches and mental status changes. Some rarely had strokes and seizures. Neurological issues can continue for years after people recover from the initial EVD infection.

Objective:

This is a natural history study to learn more about how EVD continues to affect survivors brain and nervous system after 5 years.

Eligibility:

People aged 18 years or older who participated in the PREVAIL III Neurology Substudy. Participants can be either an EVD survivor or a close contact. Close contacts are people who had a relationship with a survivor of EVD.

Design:

Participants will have 1 clinic visit.

They will have a physical exam. Their vital signs will be measured. They will also have a neurological checkup. The exam will assess their mental status. Their senses, reflexes, and coordination will be tested. They will be observed while walking to assess their gait. This exam will take about 1 hour.

Participants will have an interview. They will answer questions about any symptoms they have that may be affecting the brain or nervous system. This will take about 1 hour.

No other procedures will be performed during this visit.

DETAILED DESCRIPTION:
Study Description:

The long-term neurological sequelae of Ebola virus disease are not welldescribed. Through the PREVAIL III (PIII) Ebola Natural History Study, a Neurology Substudy was undertaken to better understand the long-term neurologic sequelae of EVD, with 5 years of follow up planned. Unfortunately, due to the COVID-19 pandemic beginning in early 2020, the final study evaluations of the PIII Neurology Substudy participants were unable to be performed by study staff based in the United States. To better understand the long-term neurological sequelae of EVD survivors, we propose this single-visit observational study of the participants of the Neurology Substudy of PIII. We hypothesize that, although the EVD survivors neurological issues have improved over time, they still may have neurological sequelae even after over 5 years convalescence from EVD.

Objectives:

Primary Objective: To characterize the neurological sequelae in EVD survivors after over 5 years convalescence from EVD

Secondary Objectives: To harmonize data from PIII Neurology substudy to determine how the prevalence of neurological complaints and neurological exam abnormalities changed over time.

Endpoints:

Primary Endpoint: The prevalence of neurological complaints and neurological exam abnormalities in EVD survivors after 5 years or more of convalescence from EVD, in comparison to close contacts.

Secondary Endpoints: The change of neurological complaints and neurological exam abnormalities in EVD survivors over time.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Male or female, aged 18 or older
3. Previous participant in the PREVAIL III Neurology Substudy, either as an EVD survivor or close contact*
4. Ability of subject to understand and the willingness to sign a written informed consent document, or indicate consent with the help of visual aids in the case of illiterate participants.

Close contacts are those who had a relationship with someone who survived EVD, but were never diagnosed with EVD themselves.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. At the time of enrollment, lacks consent capacity due to cognitive impairment that would make them incapable of understanding the explanation of the procedures in this study. Cognitive capacity to consent will be determined at the time of enrollment. Participants with mental disorders or those participants who are cognitively impaired yet still retain consent capacity will not be excluded.
2. Is unable to comply with the procedures of the protocol.
3. Has any condition in the judgement of the study staff that would make the volunteer unable to participate in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include all of the participants who were involved in the Neurology Substudy of the PREVAIL III Ebola Natural History Study who are willing to join. The Neurology Substudy originally included 172 self-identified EVD survivors and 93 self-identified close contacts. Since inclusion into the PIII study and Neurology substudy, there is bound to be some attrition (with a few participants who have passed away, some who have moved away from the area, some who simply may no longer wish to participate, among other reasons for attrition).
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
Neurological Sequelae | 5 years post initial enrollment in PREVAIL III
  To characterize the neurological sequelae in EVD survivors after over 5 years convalescence from EVD

SECONDARY OUTCOMES:
Harmonize data | 5 years post initial enrollment in PREVAIL III
  To harmonize data from PIII Neurology substudy to determine how the incidence of neurological complaints and neurological exam abnormalities changed over time

CONTACTS AND LOCATIONS:
Overall Officials: Bridgette J Billioux, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- John F. Kennedy Medical Center, Monrovia, Liberia

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share IPD that is clinically relevant and IPD that underlie results in publication.